CLINICAL TRIAL: NCT03973515
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, 4-Period, Crossover Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Three Dose Levels of the Investigational Drug (PB-201) in Drug-naive Adult Subjects With Type 2 Diabetes Mellitus as Monotherapy
Brief Title: Clinical Trial for the Investigational Drug (PB-201) in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PegBio Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PB-201
Record Dates: First submitted 2019-05-29; First posted 2019-06-04 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2019-06

CONDITIONS: Type2 Diabetes Mellitus
Keywords: Glucokinase activator(GKA); hypoglycemia
MeSH Terms: conditions — Hypoglycemia | interventions — glucokinase activator compound 50; Lead-201

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PB-201 50/50mg by mouth,every morning and noon for 7 days (Experimental)
  Interventions: Drug: glucokinase activator
- PB-201 100/50mg by mouth,every morning and noon for 7 days (Experimental)
  Interventions: Drug: glucokinase activator
- PB-201 100/100mg by mouth,every morning and noon for 7 days (Experimental)
  Interventions: Drug: glucokinase activator
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: glucokinase activator — PB-201 is a kind of dual and partial GKA
  Other Names: PB-201
  Arms: PB-201 100/100mg by mouth,every morning and noon for 7 days; PB-201 100/50mg by mouth,every morning and noon for 7 days; PB-201 50/50mg by mouth,every morning and noon for 7 days
Drug: Placebo — Placebo oral tablet
  Other Names: PB-201 Placebo
  Arms: placebo

SUMMARY:
This crossover study investigates the safety, tolerability, pharmacokinetics (PK) ,pharmacodynamics (PD) effect of three dose levels of PB-201,and characterizes the PK profile of a prominent des-methyl metabolite of PB-201(WI-0800), following dosing of three dose levels of PB-201 in drug-naive Chinese adult subjects with Type 2 diabetes mellitus (T2DM) as monotherapy.

There were 7 days separating 4 treatment periods and at least 7-day washout (but not exceeding 14 days) between dosing in 4 periods with 3 dose levels of PB-201 and placebo. Three dose levels of PB-201 are: split dose regimen of 50 mg 30 minutes before morning meal plus 50 mg 30 minutes before lunch at approximately 3.5 hours after morning dose, and split dose regimen of 100 mg 30 minutes before morning meal plus 100 mg 30 minutes before lunch at approximately 3.5 hours after morning dose, and split dose regimen of 150 mg 30 minutes before morning meal plus 100 mg 30 minutes before lunch at approximately 3.5 hours after morning dose.

ELIGIBILITY:
Inclusion Criteria:

1. Glycosylated hemoglobin (HbA1c) 7.5%-11% at screening, and 7.0%-10.0% pre-randomization
2. FPG 7.0 mmol/L-11.0mmol/L at screening and pre-randomization
3. Body mass index (BMI) 18.5 and-35.0 kg/m2 at screening
4. Antidiabetics-naive within 2 months before screening

Exclusion Criteria:

1. Diagnosis of type 1 diabetes mellitus or secondary forms of diabetes
2. History of febrile illness within 5 days prior to dosing
3. Medical history of myocardial infarction, angina/unstable angina, coronary revascularization, stroke or transient ischemic attack
4. Any medical history or current clinical evidence of congestive heart failure, New York Heart Association (NYHA) Functional Classification, Classes II-IV
5. Episode(s) of hypoglycemia adverse events (HAE) of 'severe' intensity prior to screening; either:

   1. >1 in the previous 3 months; or
   2. >2 in the previous 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Time to peak(Tmax) | 9 days
  hour
Peak Plasma Concentration (Cmax) | 9 days
  ng/mL
Area under the plasma concentration versus time curve (AUC) | 9 days
  ng•hr/mL

SECONDARY OUTCOMES:
The change for fasting plasma glucose (FPG) | 8days
  The change from baseline value (day 0) to the last dose of drug in this period (day 7) compared to placebo
The change for postprandial plasma glucose (PPG) | 8 days
  The change from baseline value (day 0) to the last dose of drug in this period (day 7) compared to placebo
The change for plasma C-peptide | 8 days
  The change from baseline value (day 0) to the last dose of drug in this period (day 7) compared to placebo
The change for plasma insulin | 8 days
  The change from baseline value (day 0) to the last dose of drug in this period (day 7) compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: HaiYan Li, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu D, Du Y, Yao X, Wei Y, Zhu J, Cui C, Zhou H, Xu M, Li H, Ji L. Safety, tolerability, pharmacokinetics, and pharmacodynamics of the glucokinase activator PB-201 and its effects on the glucose excursion profile in drug-naive Chinese patients with type 2 diabetes: a randomised controlled, crossover, single-centre phase 1 trial. EClinicalMedicine. 2021 Nov 6;42:101185. doi: 10.1016/j.eclinm.2021.101185. eCollection 2021 Dec. PMID 34805810